CLINICAL TRIAL: NCT04609241
Title: Clinical Trial for the Safety and Efficacy of Murine CD79b CAR-T Therapy for Patients With Relapsed and/or Refractory B-cell Acute Lymphoblastic Leukemia and B-cell Non-Hodgkin's Lymphoma
Brief Title: CD79b CAR-T Cell Therapy for Patients With Relapsed and/or Refractory Acute Lymphoblastic Leukemia and B-cell Non-Hodgkin's Lymphoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD79b-001
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Relapsed and/or Refractory Acute Lymphoblastic Leukemia; Relapsed and/or Refractory B-cell Non-Hodgkin's Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CD79b CAR-T Cell (Experimental)
  Interventions: Drug: CD79b CAR-T Cells

INTERVENTIONS:
Drug: CD79b CAR-T Cells — Each subject receive CD79b CAR-Tcells by intravenous infusion

SUMMARY:
A study of CD79b CAR-T Cell Therapy for Patients With Relapsed and/or Refractory Acute Lymphoblastic Leukemia and B-cell Non-Hodgkin's Lymphoma

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory Relapsed and/or Refractory Acute Lymphoblastic Leukemia and B-cell Non-Hodgkin's Lymphoma. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 72 patients will be enrolled. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

* Only For B-ALL

  1. No gender or age limit
  2. Histologically confirmed diagnosis of CD69b+ B-ALL per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Myeloid Leukemia (2016.v1);
  3. Relapsed or refractory CD123+ AML (meeting one of the following conditions):

     1. CR not achieved after standardized chemotherapy;
     2. CR achieved following the first induction, but CR duration is less than 12 months;
     3. Ineffectively after first or multiple remedial treatments;
     4. 2 or more relapses;
  4. The number of primordial cells in bone marrow is > 5% (by morphology), and/or > 0.01% (by flowcytometry);
  5. Philadelphia chromosome negative(Ph-) subjects; Ph+ subjects who cannot tolerate tyrosine kinase inhibitor (TKI) treatment or who do not respond to two kinds of TKI treatment;
* Only For B-NHL

  1. No gender or age limit;
  2. Histologically confirmed diagnosis of DLBCL (NOS), FL, DLBCL transformed from CLL/SLL, PMBCL, and HGBCL per the WHO Classification Criteria for Lymphoma (2016);
  3. Relapsed or refractory B-NHL (meeting one of the following conditions):

  <!-- -->

  1. No response or relapse after second-line or above chemotherapy regimens;
  2. Primary drug resistance;
  3. Relapse after auto-HSCT;
  4. At least one assessable tumor lesion per Lugano 2014 criteria
* For both B-ALL and B-NHL

  1. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit ofnormal, creatinine ≤ 176.8 umol/L;
  2. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%;
  3. No active infection in the lungs, blood oxygen saturation in indoorair is ≥ 92%;
  4. Estimated survival time ≥ 3 months;
  5. ECOG performance status 0 to 2;
  6. Patients or their legal guardians volunteer to participate in the studyand sign the informed consent.

Exclusion Criteria:

* 1. History of craniocerebral trauma, conscious disturbance,epilepsy,cerebrovascular ischemia, and cerebrovascular, hemorrhagicdiseases; 2. Electrocardiogram shows prolonged QT interval, severe heart diseasessuch as severe arrhythmia in the past; 3. Pregnant (or lactating) women; 4. Patients with severe active infections (excluding simple urinarytractinfectionand bacterial pharyngitis); 5. Active infection of hepatitis B virus or hepatitis C virus; 6. Previously treated with any CAR-T cell product or other genetically modified T cell therapies; 7. Insufficient amplification capacity in response to CD3 / CD28 co-stimulus signal (<5 times) 8. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl; 9. Other uncontrolled diseases that were not suitable for this trial; 10. Patients with HIV infection; 11. Any situations that the investigator believes may increase the risk ofpatients or interfere with the results of study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CD79b targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CD79b targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Acute Lymphoblastic Leukemia (ALL), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 6, 12, 18 and 24
ALL, Overall survival（OS） | Up to 2 years after CD79b CAR-T cells infusion
  From the first infusion of CD79b CAR-T cells to death or the last visit
ALL, Event-free survival (EFS) | Up to 2 years after CD79b CAR-T cells infusion
  From the first infusion of CD79b CAR-T cells to the occurrence of any event, including death, relapse or generelapse, disease progression (any one occurs first), and the last visit
B-cell Non-Hodgkin's Lymphoma（B-NHL）, Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 6, 12, 18 and 24
B-NHL, Overall survival（OS） | Up to 2 years after CD79b CAR-T cells infusion
  From the first infusion of CD79b CAR-T cells to death or the last visit
B-NHL, Event-free survival (EFS) | Up to 2 years after CD79b CAR-T cells infusion
  From the first infusion of CD79b CAR-T cells to the occurrence of any event, including death, relapse or generelapse, disease progression (any one occurs first), and the last visit
Quality of life(EORTC QLQ-C30) Core 30 (EORTC QLQ-C30) | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scores mean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Hospital Anxiety and Depression Scale (HADS) [max score: 42, min score: 0, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China